CLINICAL TRIAL: NCT00114894
Title: Field Study of the Prevention of Jellyfish Stings With a Topical Sting Inhibitor
Brief Title: Prevention of Jellyfish Stings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0311M54041
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Bites and Stings
Keywords: Jellyfish; Stings; Marine; Envenomation; Jellyfish stings
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safe Sea (Experimental)
  Interventions: Other: Safe Sea ™
- Placebo (Sham Comparator): Coppertone® SPF15 (Schering-Plough)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Safe Sea ™ — Safe Sea ™ applied one time at 2 mg/cm2 coverage
  Arms: Safe Sea
Other: Placebo — Placebo Coppertone® SPF15 sunscreen(Schering-Plough) applied at 2 mg/cm2 body coverage
  Arms: Placebo

SUMMARY:
Jellyfish stings are a common occurrence among ocean-goers worldwide with an estimated 150 million envenomations annually. Fatalities and hospitalizations occur annually, particularly in the Indo-Pacific regions. A new topical jellyfish sting inhibitor based on the mucous coating of the clown fish prevents 85% of jellyfish stings in laboratory settings. The field effectiveness is unknown. This is a field test to determine the real world effectiveness.

DETAILED DESCRIPTION:
Jellyfish stings are a common occurrence among ocean-goers worldwide with an estimated 150 million envenomations annually. Fatalities and hospitalizations occur annually, particularly in the Indo-Pacific regions. A new topical jellyfish sting inhibitor based on the mucous coating of the clown fish prevents 85% of jellyfish stings in laboratory settings.

Clown fish inhabit within the tentacles of sea anemones, which have stinging cells similar to those of jellyfish, yet clown fish are not stung by the sea anemones. In controlled laboratory environments, the jellyfish sting inhibitor, Safe Sea™ when applied to volunteers' arms, prevented 100% of Chrysaora fuscescens stings and 70% of Chiropsalmus quadrumanus stings. Of the C. quadrumanus stings that occurred, their intensity was diminished. The field effectiveness is unknown. This is a field test to determine the real world effectiveness of Safe Sea to prevent jellyfish stings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers planning on snorkeling for 30 to 45 minutes.

Exclusion Criteria:

* Pregnancy
* Severe allergy to jellyfish
* Allergy to any topical dermatologic product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-04; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Incidence of jellyfish stings | during recreational saltwater exposure (~30 min)

SECONDARY OUTCOMES:
Occurrence of seabather's eruption | within 48 hours of saltwater exposure
impact of body hair on jellyfish stings | after recreational saltwater exposure

CONTACTS AND LOCATIONS:
Overall Officials: David R Boulware, MD, Principal Investigator — University of Minnesota
Locations (1):
- Dry Tortugas National Park, Key West, Florida, United States

REFERENCES:
- [Result] Boulware DR. A randomized, controlled field trial for the prevention of jellyfish stings with a topical sting inhibitor. J Travel Med. 2006 May-Jun;13(3):166-71. doi: 10.1111/j.1708-8305.2006.00036.x. PMID 16706948